CLINICAL TRIAL: NCT04132414
Title: Monitoring Of REgional Cerebral Oxygenation (rcSO2 ) With Near INFrared SpectrOscopy (NIRS) During Non-cardiac Surgery in Preterms, Neonates and Infants in Addition to Standard Monitoring to Guide Intraoperative Management
Brief Title: Cerebral NIRS Monitoring During Anesthesia in Neonates and Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study investigators changed institution
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 31-175 ex 18/19
Record Dates: First submitted 2019-09-05; First posted 2019-10-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Oxygenation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NIRS open (Experimental): Cerebral NIRS monitoring applied and visible to caregiver. Interventions according to protocol in phases of cerebral hypoxia
  Interventions: Diagnostic Test: NIRS open
- NIRS blinded (No Intervention): NIRS monitoring applied and masked for caregiver.

INTERVENTIONS:
Diagnostic Test: NIRS open — Treatment according to protocol in phases of cerebral hypoxia.
  Arms: NIRS open

SUMMARY:
The brain is a very vulnerable organ, especially in premature babies, newborns and infants. However, during anesthesia, the oxygenation of the brain can only be monitored indirectly and insufficiently. Near-infrared spectroscopy (NIRS) is an established monitoring method in other areas (e.g., neonatology, cardiac anesthesia), which provides non-invasive information about the regional oxygen supply of the brain. The integration of this monitoring device into the anaesthesiological care for neonates and infants could reduce the risk of cerebral hypoxia. The planned study investigates whether the use of NIRS in anesthetized children up to 6 months can prevent or influence the occurrence of cerebral hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Expected duration of Anesthesia >45 minutes
* Intervention/surgery in the operating room

Exclusion Criteria:

* Impossibility to place cerebral NIRS sensor
* Known cerebral pathology
* Missing parental consent
* Congenial cardiac condition with right to left shunt
* Cardiac surgery

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral hypoxic burden | 1 day
  Time under 65% cerebral oxygen saturation

SECONDARY OUTCOMES:
Fluid administration | 1 day
  ml/kg
Number of participants with Vasopressor or Inotrope administered | 1 day
  Proportion
Number of participants with erythrocyte administration | 1 day
  Proportion
Fraction of inspired oxygen | 1 day
  %

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Heschl, M.D., Ph.D., Principal Investigator — Medical University of Graz

IPD SHARING:
Plan to Share IPD: No